CLINICAL TRIAL: NCT07178938
Title: An International, Multicenter, Open-label, Multicohort, Platform Trial Assessing Uptake, Safety and Efficacy of Theranostic Agents in Solid Tumors With Active Brain Metastases (the THERANOVA Study; NMN-02).
Brief Title: Platform Trial Assessing Uptake, Safety and Efficacy of Theranostic Agents in Solid Tumors With Active Brain Metastases
Acronym: THERANOVA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEDOPP838
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors; HER2-positive Breast Cancer
Keywords: THERANOVA; Platform trial; Active Brain Metastases; Theranostic Agents; Radioligand therapy; Radioligand imaging
MeSH Terms: interventions — somatostatin receptor 2

STUDY DESIGN:
Intervention Model Description: An international, multicenter, open-label, multicohort, platform trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: Radiotracer targeting somatostatin receptor 2 (SSTR2) ([68Ga]Ga-DOTA-TOC)

INTERVENTIONS:
Drug: Radiotracer targeting somatostatin receptor 2 (SSTR2) ([68Ga]Ga-DOTA-TOC) — Patients will receive a single infusion of the diagnostic agent [68Ga]Ga-DOTA-TOC will which will be detected by Positron Emission Tomography/Computed Tomography (PET/CT) imaging. The recommended activity for an adult weighing 70 kg is 100 to 200 MBq, administered by direct slow intravenous injection and for a single use only.

SUMMARY:
This trial will evaluate treatment for patients with solid tumors with active brain metastases. Patients will be treated with a theranostic or diagnostic agent. Theranostic agents are targeted radioactive drugs used to identify (diagnose) and to deliver therapy. The main purpose of the study is to analyze the efficacy (to find out how effective a treatment is) of each of the theranostic agents in patients who have solid tumors with active brain metastases. In the diagnostic phase, the main objective is to determine the proportion of patients showing target expression in the brain lesion after a single dose of diagnostic agent. In the therapeutic phase, the theranostic agent's efficacy will be determined by assessing the response rate in the brain, defined as intracranial response rate at 24 weeks.

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, multicohort, platform design trial comprising the development of theranostic cards, and diagnostic and therapeutic phases.

Based on the preliminary analysis, the platform identifies the best strategy for the clinical development of each specific Investigational Medicinal Product (IMP) in the context of solid tumors and active brain metastases. The flexible design of the trial adapts to the specific developmental needs of each IMP. Analysis of each agent will be performed extracting preliminary data from available sources and literature review.

The diagnostic phase is comprised of three Stages. The therapeutic phase is comprised of two Stages.

Patients enrolled must be ≥18 years of age with solid tumors and active brain metastases (BMs), who have evidence of at least one measurable brain lesion of ≥10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging (MRI) according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, life expectancy ≥ 6 weeks, and adequate bone marrow and organ function are mandatory.

After treatment discontinuation (EoT), all patients will have a safety visit scheduled 28 days (± 7 days) after the last dose of IMP, in order to follow up toxicities and changes in concomitant medication. Should alternative timelines be necessary based on the IMP, these will be detailed in the corresponding appendix. After the safety visit, all patients treated in the therapeutic phase will enter a post treatment follow-up period during which survival status and subsequent anticancer therapy information will be collected every 3 months (± 7 days) until death, lost to follow-up, elective withdrawal from the study, or the End of Study (EoS), whichever occurs first. This information may be collected by telephone call. Patients who discontinue treatment without evidence of disease progression will be followed every 6 months (± 14 days) for tumor assessments until documented progression, elective withdrawal from the study, the start of new anti-cancer treatment, or study completion or termination.

Safety long-term follow-up will be established based on the cohort and the specific IMP as explained in the IMP specific appendix section.

The THERANOVA Expert Committee took the decision to test the radiotracer targeting somatostatin receptor 2 (SSTR2) ([68Ga]Ga-DOTA-TOC) in the diagnostic phase for patients with Human Epidermal Growth Factor Receptor (HER2)-positive breast cancer and brain metastases as the first cohort. The decision to assess [68Ga]Ga-DOTA-TOC in the diagnostic phase for this population reflects the potential of Radioligand therapies (RLTs) to target brain lesions. The current platform Study incorporates essential design components that may be crucial for a comprehensive evaluation of the balance between benefits and risks of [68Ga]Ga-DOTA-TOC in patients with solid tumors and BMs. The eligibility criteria are designed to maximize the diagnostic value of [68Ga]Ga-DOTA-TOC and minimize its potential associated risks.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this trial, an individual must meet ALL the following criteria:

1. Patient, or legal representative (if applicable), must be capable to understand the purpose of the study and have signed written Informed Consent Form (ICF) prior to beginning specific protocol procedures.
2. Male or female patients ≥ 18 years of age at the time of signing ICF.
3. Radiologically documented locally advanced unresectable or metastatic breast cancer (BC).
4. Histologically confirmed HER2-positive (HER2[+]) breast cancer based on local testing on the most recent analyzed biopsy according to the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
5. Untreated newly diagnosed or progressing brain metastasis (BM) after prior local therapy. Any number of brain lesions is acceptable as long as all the eligibility criteria are fulfilled.
6. Measurable disease according to Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria, with at least one measurable brain lesion of ≥ 10 mm on T1-weighted, gadolinium-enhanced magnetic resonance imaging (MRI).
7. Patients may or may not have type I leptomeningeal disease (LMD) per European Association of Neuro-Oncology (EANO)- European Society for Molecular Oncology (ESMO) criteria.
8. Stable or decreasing corticosteroid dose, or no use of corticoids, for at least 7 days prior to enrollment.
9. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 2.
10. Minimum life expectancy of ≥ 6 weeks at screening.
11. Resolution of all acute toxic effects of prior anticancer therapy to grade ≤ 1 as determined by the US National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (v.5.0).

    Note: except for alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion.
12. Patient has adequate bone marrow, liver, and renal function within 7 days before first Study treatment dose:

    I. Hematological (without platelet, red blood cell transfusion/plasma transfusion within 1 week prior to screening assessment, and/or granulocyte colony-stimulating factor support): White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 9.0 g/dL (≥ 5.6 mmol/L).

    II. Hepatic: Serum albumin ≥ 2.5 g/dL; total bilirubin ≤ 1.5 times upper limit of normal (ULN) (≤ 3 in patients with liver metastases or know history of Gilbert's disease); alkaline phosphatase (ALP) ≤ 2.5 times ULN (≤ 5 in patients with liver metastases); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times ULN (≤ 5 in patients with liver metastases); international normalized ratio (INR) < 1.5.

    III. Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 based on Cockcroft-Gault glomerular filtration rate estimation for patients with creatinine levels above institutional normal.
13. Women of childbearing potential who are sexually active with a non-sterilized male partner must have a negative serum pregnancy test within 14 days before Study treatment initiation. In addition, they must agree to use one highly effective method of birth control for the full duration of study participation.
14. Male participants who are sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception for the full duration of study participation.
15. Patients must be accessible for treatment and follow-up.

Exclusion Criteria

An individual who meets ANY of the following criteria will be excluded from participation in this trial:

1. Participation in another clinical trial, interventional or observational, until the Study's safety visit (participation in retrospective studies or data analysis is allowed).
2. Treatment with approved or investigational cancer therapy within 14 days prior to initiation of study drug.
3. Known history of invasive malignancy and other than the malignancy of interest within 5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. For other cancers considered to have a low risk of recurrence, discussion with the Sponsor's Medical Monitor is required.
4. Known allergy or hypersensitivity reaction to any investigational medicinal products (diagnostic radioligand) or their incorporated substances.
5. Major surgical procedure or significant traumatic injury within 14 days before the first dose of study treatment or anticipation of need for major surgery within the course of the study treatment.
6. Pregnant or breastfeeding females or patients not willing to apply highly effective contraception as defined in the protocol.
7. Receipt of live or attenuated vaccine within 30 days prior to the first dose of study treatment.
8. Has active or uncontrolled infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
9. Has known human immunodeficiency virus (HIV) infection that is not well controlled.
10. Other active uncontrolled infection at the time of enrollment.
11. Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
12. A history of uncontrolled seizures, central nervous system (CNS) disorders, or serious and/or unstable pre-existing psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs or interfering with trial participant safety.
13. Known substance abuse or any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation.
14. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study.
15. Inability or unwillingness to comply with the requirements of the protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients showing target expression | Up to two months
  Proportion of patients showing target expression (Maximum Standardized Uptake Value (SUVmax) equal to or greater than 2.3) in brain lesion as measured by PET/CT.

SECONDARY OUTCOMES:
Percentage of intracranial (IC) lesions | Up to two months
  Percentage of IC lesions showing PET/CT targeted expression (SUVmax equal to or greater than 2.3).
Percentage of extracranial (EC) lesions | Up tp two months
  Percentage of EC lesions showing PET/CT targeted expression (SUVmax equal to or greater than 2.3).
Maximum standardized uptake value | Up to two months
  The maximum standardized uptake value (SUVmax and Mean Standardized Uptake Value (SUVmean)) in brain lesions and their relative values compared to normal liver and blood pool activity.
Incidence of Diagnostic radioligand-Emergent Adverse Events (Safety and tolerability) | Up to two months
  Determine the safety and toxicity profile of the selected diagnostic radioligand in patients with advanced solid tumors and active BMs according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0).
Incidence of Diagnostic Radioligand-Emergent Adverse Events, Serious Adverse Events and Suspected Unexpected Serious Adverse Reactions | Up to two months
  Determine the safety and toxicity profile of the selected diagnostic radioligand in patients with advanced solid tumors and active BMs according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0) (Safety and Tolerability)

IPD SHARING:
Plan to Share IPD: Yes
Data collected within this study will be made available to researchers after contacting the corresponding author and upon revision and approval based on scientific merit by the trial management group (which includes a qualified statistician) of a detailed proposal for their use. The data required for the approved, specified purposes and the trial protocol will be provided after the completion of a data-sharing agreement that will be set up by the study sponsor. All data provided are anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. Data sharing should begin 1 month after publication of study main results and ending 5 years after article publication. Estimate timeframe for response will be within 30 days.